CLINICAL TRIAL: NCT03558126
Title: Silicone Tube Miniature Drainage Device Implanted Under Scleral Flap for the Surgical Treatment of Glaucoma
Brief Title: Silicone Tube for the Surgical Treatment of Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: yin ying zhao (Other)
Responsible Party: Sponsor-Investigator, yin ying zhao, Zhejiang Eye Hospital, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL-HZ-tube
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Glaucoma, Open-Angle
Keywords: silicone tube; miniature drainage device; POAG; IOP
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: silicone tube

SUMMARY:
The biocompatible silicone tube miniature drainage device is a small, non-valved implant to shunt aqueous humor underneath the conjunctiva to control the intraocular pressure. Efficacy and safety were evaluated with a minimum follow-up of 12 months.

DETAILED DESCRIPTION:
Patients were examined postoperatively at 1 day, 1 week, 1, 3, 6, 12, 18, 24 months or more frequent when required. IOP, BCVA and slit lamp biomicroscopy were observed at every visit. History of all medication details and postoperative complications were recorded. One-way analysis of variance (ANOVA) with repeated measures was used to analyze the other differences over time in IOP and BCVA. Nonparametric K-related samples test was used to analyze the difference of medications number at different time points. Success rates were evaluated using Kaplan-Meyer survival analysis curves.

ELIGIBILITY:
Inclusion Criteria:Eligible patients were at least 18 years of age and presented with medically uncontrolled POAG requiring incisional surgery for IOP (intraocular pressure) reduction.

-

Exclusion Criteria:Exclusion criteria included narrow angles, normal tension glaucoma, previous eye surgery (except cataract surgery), neovascular glaucoma, uveitis, any ocular abnormality that would preclude accurate IOP assessment, and inability to comply with the follow-up program or unwillingness to participate in this study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
IOP | 3 years
  Intraocular pressure

SECONDARY OUTCOMES:
Number of anti-glaucoma medication | 3 years
  Number of anti-glaucoma medication

IPD SHARING:
Plan to Share IPD: No